CLINICAL TRIAL: NCT03034863
Title: SAFER: A Brief Intervention Involving Family Members in Suicide Safety Planning
Acronym: SAFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2432-R; RX002432-01 (Other Grant/Funding Number: VA ORD)
Record Dates: First submitted 2017-01-11; First posted 2017-01-27 (Estimated); Results first posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-11

CONDITIONS: Suicide
Keywords: Family Caregivers; Spouse Caregivers; Veterans; Suicide; Clinical Trial; Military Families; Military Psychology
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The individual who evaluates the outcomes of interest will not know the assigned condition of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SAFER (Experimental): SAFER (Safe Actions for Families to Encourage Recovery): A novel, 5-session intervention to enhance currently mandated VA suicide safety planning by involving supporting partners to support its implementation. Incorporation of education about suicide risk factors and teaching communication skills of active listening and making a positive request will supply Veterans and supporting partners with the knowledge and tools needed to 1) identify potential warning signs, and 2) discuss Veteran ideation or partner concerns with assurance that such requests will be listened to with validation and support, creating an ally for the suicidal Veteran in his struggle. As discussed above, research has demonstrated compellingly that suicidal desire is motivated by two interpersonal factors; perceived burdensomeness and thwarted belongingness. SAFER aims to increase partner support for the Veteran to directly mitigate Veteran loneliness and sense of being a burden to others.
  Interventions: Behavioral: Safe Actions for Families to Encourage Recovery
- I-SPI (Active Comparator): The comparison condition will be an assessment-only enhanced treatment-as-usual called the Individual Safety Planning Intervention (I-SPI), incorporating weekly scripted check-in phone calls to review mood symptoms and use of the safety plan, which will then be given as feedback to the Veteran's primary mental health provider.
  Interventions: Behavioral: Individual Safety Planning Intervention

INTERVENTIONS:
Behavioral: Safe Actions for Families to Encourage Recovery — A novel, 5-session intervention to enhance currently mandated VA suicide safety planning by involving family members to support its implementation. Incorporation of education about suicide risk factors and teaching communication skills of active listening and making a positive request will supply Veterans and family members with the knowledge and tools needed to 1) identify potential warning signs, and 2) discuss Veteran ideation or family concerns with assurance that such requests will be listened to with validation and support, creating an ally for the suicidal Veteran in his struggle. As discussed above, research has demonstrated compellingly that suicidal desire is motivated by two interpersonal factors; perceived burdensomeness and thwarted belongingness. SAFER aims to increase family support for the Veteran to directly mitigate Veteran loneliness and sense of being a burden to others.
  Other Names: SAFER
  Arms: SAFER
Behavioral: Individual Safety Planning Intervention — The comparison condition will be an assessment-only enhanced treatment-as-usual intervention called the Individual Safety Planning Intervention (I-SPI).
  Other Names: I-SPI
  Arms: I-SPI

SUMMARY:
The management of suicide risk is a pressing national public health issue especially among Veterans, and there exist no guidelines of how best to involve family members in this effort. This proposal will integrate family and couples communication skills training with suicide safety planning. The goal is for the sharing of Veteran suicide safety plans with family members and the construction of a parallel family member safety plan, in efforts to mobilize and support family involvement.

DETAILED DESCRIPTION:
Psychological models of suicidality emphasize the role of social factors in the development and intensification of suicidal thoughts and behavior, including feeling like a burden on family and friends, feelings of isolation and not belonging, and perceptions of diminished support from one's family and social network. Despite the critical role of family factors in protecting against suicidality, families lack education on how their behavior can help avert or unwittingly aggravate suicidal thoughts/ behavior. Families worry about their relative but feel uncertain of how to help and need professional guidance. Family worries about suicidality are associated with compromised family physical and mental health and consequently, diminished ability to offer needed support. Because suicide safety plans rely on mobilizing support in times of crisis, families need to be equipped to provide needed support.

Family recommendations from the VA Behavioral Health Autopsy Program (BHAP) Annual Report 6/30/15 based on interviews with 114 family members highlighted the importance of:

1. educating families about suicide warning signs:
2. improving communication between the veteran and family member
3. involving the family in the veterans' treatment to enhance support and trust
4. providing families with coaching on how to assist their loved one to seek help.

Management of suicidal behavior is covered in comprehensive family psychoeducation programs, but there is an urgent need for a brief family-based intervention specifically focused on suicide prevention that can be used in conjunction with the currently mandated SSP and as a part of routine care.

Despite the enrichment of VA suicide prevention services and implementation of the national suicide hotline, Veteran suicide completions have risen to 22 per day and suicide attempts numbered over 15,000 in 2012. These data underscore the urgency of developing additional interventions targeting suicidal Veterans. One potential avenue to further suicide treatment and rehabilitation efforts is to develop strategies that maximize family support, however almost no family interventions exist for suicidal Veterans. The construction of a Suicide Safety Plan (SSP); a "best practice," is mandated throughout the VA system, and a vital component of the VA's coordinated effort at suicide prevention and recovery. The pilot data on patterns of SSP use in suicidal Veterans highlighted the importance of sharing the plan with family or close friends. However, respondents also noted significant obstacles in their ability to reach out to others when in distress. To the knowledge of Investigators, there are currently no recommended guidelines or mechanisms for involving family in safety planning, despite its inclusion as a step of the plan. "Safe Actions for Families to Encourage Recovery" (SAFER) a novel suicide safety planning family intervention has been designed to fill this critical gap and provide a mechanism to communicate about safety planning. SAFER, a 4-session, family intervention, combines education about suicide and suicide safety planning with communication skills training from evidence-based practices. The aim is to facilitate communication about suicide safety planning and to develop both a Veteran and family member safety plan.

Data from this project will test the intervention's feasibility, acceptability and preliminary efficacy in a Stage II small-scale randomized clinical trial in 39 moderate suicide risk Veterans and their supporting partners. The comparison condition will be safety planning without supporting partner involvement plus weekly check-in phone calls. Primary Veteran outcomes include reducing suicidal ideation/behavior. Secondary Veteran outcomes include reducing suicidal cognitions (hopelessness, perceived burdensomeness, thwarted belongingness) and depression and improving subjective social support. Supporting Partner primary outcomes include reducing caregiver burden and secondary outcomes of improving suicide-related coping and family empowerment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria-Veterans:

* Eligible Veterans must be identified as at moderate risk for suicide, defined as:

  * evidence of current (within the past week) suicidal ideation
  * plan or intent on the Columbia Suicide Severity Rating Scale (C-SSRS), but scoring less than or equal to 4 on the C-SSRS Behavior Scale, and without history of a lethal suicide attempt in the last 3 months.

Inclusion criteria also include the availability of a consenting, qualifying family member or spouse/cohabiting partner.

Inclusion criteria-family member/significant others:

* Family members/friends must meet at least three (two for nonrelatives) of five criteria:

  * is a spouse, co-habiting significant other or parent
  * has more frequent contact than any other caregiver
  * helps to support the patient financially
  * is contacted by treatment staff for emergencies
  * has been involved in the patient's treatment

Exclusion Criteria:

Exclusion criteria for Veterans and family/partners are:

* untreated or un-medicated psychosis
* current alcohol or drug abuse or dependence defined by a Patient Health Questionnaire (PHQ) for Alcohol & Drug Use
* for couples, "severe" intimate-partner violence as defined by the revised 20-item Conflict Tactics Scale Short Form (CTS2S)
* medical condition or life event, e.g.,
* participation in another family-based psychosocial intervention trial six months prior to study
* limited English proficiency. Participants will be screened for inclusion/exclusion as described above immediately after giving consent.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne S. Goodman, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited, consented, and randomized 39 Veterans at risk for suicide and 39 corresponding supporting partners over a 30-month period from a large VA medical center in a major metropolitan area in the North East. Recruitment sources included VA suicide prevention coordinators, a Veteran's primary clinician from the VA Medical Center's (VAMC) psychiatric inpatient unit or outpatient care center, or through community outreach (e.g., Vet Centers and higher education institutions).
Groups:
- SAFER: Safe Actions for Families to Encourage Recovery (SAFER): A novel, 4-session intervention to enhance currently mandated VA suicide safety planning by involving family members to support its implementation. Incorporation of education about suicide risk factors and teaching communication skills of active listening and making a positive request will supply Veterans and family members with the knowledge and tools needed to 1) identify potential warning signs, and 2) discuss Veteran ideation or family concerns. SAFER aims to increase family support for the Veteran to directly mitigate Veteran loneliness and sense of being a burden to others.
  Safe Actions for Families to Encourage Recovery: A novel, 4-session intervention to enhance VA suicide safety planning by involving family members to support its implementation.
- I-SPI: The comparison condition will be an assessment-only enhanced treatment-as-usual, the currently mandated Individual Safety Planning Intervention (I-SPI). I-SPI incorporates update and use of the safety plan, which will then be uploaded to the Computerized Patient Record System (CPRS) so the Veterans' primary mental health providers can access.
  Treatment-as-Usual: The comparison condition will be an assessment-only enhanced treatment-as-usual called the Individual Safety Planning Intervention (I-SPI).
Period: Overall Study
Arm/Group | SAFER | I-SPI
Started | 38 | 40
Veterans | 19 | 20
Supporting Partners | 19 | 20
Completed | 28 | 28
Not Completed | 10 | 12

BASELINE CHARACTERISTICS:
Population: The overall sample included 39 veterans with recent suicidal ideation and/or a history of a suicide attempt. The 39 dyads also included a variety of relationships including 14 romantic partners, 13 non-romantic family members (e.g., adult children of veterans, veterans' parents), and 12 close friends.
Groups:
- SAFER: SAFER: A novel, 4-session intervention to enhance currently mandated VA suicide safety planning by involving family members to support its implementation. Incorporation of education about suicide risk factors and teaching communication skills of active listening and making a positive request will supply Veterans and family members with the knowledge and tools needed to 1) identify potential warning signs, and 2) discuss Veteran ideation or family concerns with assurance that such requests will be listened to with validation and support, creating an ally for the suicidal Veteran in his struggle. As discussed above, research has demonstrated compellingly that suicidal desire is motivated by two interpersonal factors; perceived burdensomeness and thwarted belongingness. SAFER aims to increase family support for the Veteran to directly mitigate Veteran loneliness and sense of being a burden to others.
  Safe Actions for Families to Encourage Recovery: A novel, 4-session intervention to enhance currently mandated VA suicide safety planning by involving family members to support its implementation.
- I-SPI: The comparison condition will be an assessment-only enhanced treatment-as-usual (E-TAU), the currently mandated Individual Safety Planning Intervention (I-SPI). I-SPI incorporates weekly scripted check-in phone calls to review mood symptoms and use of the safety plan, which will then be given as feedback to the Veteran's primary mental health provider.
  Treatment-as-Usual: The comparison condition will be an assessment-only enhanced treatment-as-usual called the Individual Safety Planning Intervention (I-SPI).
- Total: Total of all reporting groups
Arm/Group | SAFER | I-SPI | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Categorical [Count of Participants; unit: Participants] — This baseline measure specifically looks at Veterans. Population: Number analyzed in row differs from overall because this specifically looked at Veteran age whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 18 | 17 | 35
    >=65 years | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants] — This baseline measure specifically looks at caregivers. Population: Number analyzed in row differs from overall because this specifically looked at caregiver age whereas overall number includes both caregiver and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    <=18 years | 1 | 0 | 1
    Between 18 and 65 years | 15 | 19 | 34
    >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] — This baseline measure specifically looks at Veterans. Population: Number analyzed in row differs from overall because this specifically looked at Veteran age whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  years
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 53.26 (12.37) | 51.90 (15.62) | 52.58 (14.00)
Age, Continuous [Mean (Standard Deviation); unit: years] — This baseline measure specifically looks at caregivers. Population: Number analyzed in row differs from overall because this specifically looked at caregiver age whereas overall number includes both caregiver and their dyad partner. Therefore the number analyzed is half the total of each condition.
  years
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 48.68 (16.24) | 42.55 (12.80) | 45.62 (14.52)
Sex: Female, Male [Count of Participants; unit: Participants] — This baseline measure specifically looks at Veterans. Population: Number analyzed in row differs from overall because this specifically looked at Veteran sex whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    Female | 2 | 4 | 6
    Male | 17 | 16 | 33
Sex: Female, Male [Count of Participants; unit: Participants] — This baseline measure specifically looks at caregivers. Population: Number analyzed in row differs from overall because this specifically looked at caregiver sex whereas overall number includes both caregiver and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    Female | 13 | 12 | 25
    Male | 6 | 8 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — This baseline measure specifically looks at Veterans. Population: Number analyzed in row differs from overall because this specifically looked at Veteran ethnicity whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    Hispanic or Latino | 5 | 8 | 13
    Not Hispanic or Latino | 14 | 11 | 25
    Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — This baseline measure specifically looks at caregivers. Population: Number analyzed in row differs from overall because this specifically looked at caregiver ethnicity whereas overall number includes both caregiver and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    Hispanic or Latino | 6 | 8 | 14
    Not Hispanic or Latino | 13 | 12 | 25
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — This baseline measure specifically looks at Veterans. Population: Number analyzed in row differs from overall because this specifically looked at Veteran race whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 10 | 10 | 20
    White | 5 | 2 | 7
    More than one race | 2 | 4 | 6
    Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — This baseline measure specifically looks at caregivers. Population: Number analyzed in row differs from overall because this specifically looked at caregiver race whereas overall number includes both caregiver and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    American Indian or Alaska Native | 1 | 1 | 2
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 8 | 10 | 18
    White | 5 | 2 | 7
    More than one race | 1 | 4 | 5
    Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants] — This baseline measure specifically looks at Veterans. Population: Number analyzed in row differs from overall because this specifically looked at Veteran region of enrollment whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    United States: number analyzed (Participants) | 19 | 20 | 39
    United States | 19 | 20 | 39
Region of Enrollment [Count of Participants; unit: Participants] — This baseline measure specifically looks at caregivers. Population: Number analyzed in row differs from overall because this specifically looked at caregiver region of enrollment whereas overall number includes both caregiver and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    United States: number analyzed (Participants) | 19 | 20 | 39
    United States | 19 | 20 | 39
Veteran Suicidal Ideation [Mean (Standard Deviation); unit: units on a scale] — Moderate suicidality was measured to determine eligibility using the Columbia Suicide Severity Rating Scale (C-SSRS). The psychometric properties of the C-SSRS across multiple studies suggest moderate to strong validity and internal consistency of the ideation intensity subscale (Cronbach's alpha 0.73-0.946; Posner et al., 2011). The baseline C-SSRS measured recent (past 3 months) and lifetime severity of suicidal ideation. Baseline ideation scores were based on recent ideation. Scores range from 0 to 5. High scores mean a worse outcome (more severe ideation). Population: Number analyzed in row differs from overall because this specifically looked at Veteran suicidal ideation whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 3.26 (1.69) | 3.75 (1.33) | 3.51 (1.51)
Veteran Suicide-Related Coping [Mean (Standard Deviation); unit: units on a scale] — Suicide-related coping was evaluated by the Suicide-related Coping Scale (SRCS), a 17-item self-report measure assessing one's ability to cope with suicidal ideation and urges (Stanley, Green, Ghahramanlou-Holloway, Brenner, & Brown, 2017). The scale demonstrated good internal consistency (α=.85) at baseline; scores were averaged so that higher scores represent greater confidence and breadth of approaches to coping with suicidal thoughts and feelings (better outcome). SRCS scores have a minimum of 0 and a maximum of 4. Population: Number analyzed in row differs from overall because this specifically looked at Veteran suicide-related coping whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 3.03 (0.71) | 2.91 (0.65) | 2.97 (0.68)
Partner Support of Suicide-Related Coping [Mean (Standard Deviation); unit: units on a scale] — Supporting partners also completed five items adapted from the SRCS that assessed their confidence in their ability to support the Veteran through their suicidal urges. Items were rated on a 0 (Strongly Disagree) to 4 (Strongly Agree) scale and were averaged with higher scores indicating greater self-efficacy when supporting the Veteran through suicidal crises (better outcome). In addition to face validity, the scale showed acceptable internal consistency in the sample (α=.78). Partner SRCS scores range from 0 (minimum) to 4 (maximum). Population: Number analyzed in row differs from overall because this specifically looked at Partner support of suicide-related coping whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 3.23 (0.81) | 3.37 (0.87) | 3.3 (0.84)
Veteran Thwarted Belongingness [Mean (Standard Deviation); unit: units on a scale] — Thwarted belongingness was evaluated by the Interpersonal Needs Questionnaire (INQ-15; Van Orden, Cukrowicz, Witte, & Joiner, 2012). Scores on each subscale were averaged so that higher scores represent a greater degree of their respective constructs. Thwarted Belongingness showed acceptable internal consistency in this sample (α =.79). Thwarted belongingness scores range from 1 (minimum) to 6 (maximum). Higher scores mean a worse outcome (decreased feelings of belongingness). Population: Number analyzed in row differs from overall because this specifically looked at Veteran thwarted belongingness whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 3.23 (1.02) | 3.62 (0.9) | 3.43 (0.96)
Veteran Perceived Burdensomeness [Mean (Standard Deviation); unit: units on a scale] — Perceived burdensomeness was evaluated by the Interpersonal Needs Questionnaire (INQ-15; Van Orden, Cukrowicz, Witte, & Joiner, 2012). Scores on each subscale were averaged so that higher scores represent a greater degree of their respective constructs. Perceived Burdensomeness demonstrated excellent internal consistency in this sample (α= .95). Perceived burdensomeness scores range from 1 (minimum) to 6 (maximum). Higher scores mean a worse outcome (greater perceived burdensomeness). Population: Number analyzed in row differs from overall because this specifically looked at Veteran perceived burdensomeness whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 2.84 (1.56) | 3.03 (1.61) | 2.94 (1.59)
Supporting Partner Caregiver Burden [Mean (Standard Deviation); unit: units on a scale] — Caregiver burden was evaluated using the Caregiver Burden Inventory (CBI; Novak & Guest, 1989), a 24-item scale assessing caregiver burden in five areas: time, physical, social, developmental, and emotional burden. Items were averaged to create an overall measure of caregiver burden and showed excellent internal consistency in this study (α =.94). CBI scores range from 0 (minimum) to 4 (maximum). Higher scores mean a worse outcome (greater caregiver burden). Population: Number analyzed in row differs from overall because this specifically looked at Partner caregiver burden whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 1.39 (0.92) | 1.06 (0.96) | 1.23 (0.94)
Veteran Hopelessness [Mean (Standard Deviation); unit: units on a scale] — Veteran hopelessness will be evaluated by the Beck Hopelessness Scale (BHS), a 20-item self-report measure with adequate reliability and validity which has been predictive of suicide in psychiatric inpatients. The BHS measures three aspects of hopelessness: feelings about the future, loss of motivation, and expectations. Items are true-false and are summed to get a total BHS score, ranging from 0 to 20. Higher scores reflect a worse outcome (greater hopelessness). Population: Number analyzed in row differs from overall because this specifically looked at Veteran hopelessness whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 6.95 (5.79) | 11.72 (6.57) | 9.34 (6.18)
Veteran Depression [Mean (Standard Deviation); unit: units on a scale] — Veteran depression will be evaluated by the widely-used Beck Depression Inventory-II (BDI-II) (Cronbach's = .92). The BDI-II contains 21 items assessing depressive symptoms, each with minimum scores of 0 and maximum scores of 3. Item scores were summed, leading to a total score range of 0-63. Higher scores mean a worse outcome (more severe depressive symptoms). Population: Number analyzed in row differs from overall because this specifically looked at Veteran depression whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 24.36 (11.75) | 32.5 (15.56) | 28.43 (13.66)
Caregiver's Empowerment to Help Veteran [Mean (Standard Deviation); unit: units on a scale] — Caregiving self-efficacy/empowerment will be evaluated using the 12-item family subscale from the Family Empowerment Scale. This scale assesses the family's knowledge of mental health services and perceived ability to manage crises, and has demonstrated sensitivity to change in family intervention studies. Each item has a minimum score of 1 and a maximum score of 5, and were averaged to create a total score range of 1-5. Higher scores mean a better outcome (greater empowerment). Population: Number analyzed in row differs from overall because this specifically looked at Partner caregiver empowerment whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 3.79 (0.64) | 3.75 (0.80) | 3.77 (0.72)
Veteran's Report of Family Problem Solving [Mean (Standard Deviation); unit: units on a scale] — Veterans' reports of family problem solving will be evaluated by the 5-item Problem Solving subscale of the Family Assessment Device (FAD). Subscales have acceptable internal consistency (α = .72 to .83). Each item has a minimum score of 1 and a maximum score of 4, and were averaged to create a total score range of 1-4. Higher scores reflect worse outcomes (lower problem solving ability). Population: Number analyzed in row differs from overall because this specifically looked at Veteran reports of family problem solving whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 2.27 (0.62) | 2.44 (0.74) | 2.36 (0.68)
Veteran's Reports of Family Communication [Mean (Standard Deviation); unit: units on a scale] — Veterans' reports of family communication will be evaluated by the 6-item Communication subscale of the Family Assessment Device (FAD). Subscales have acceptable internal consistency (α = .72 to .83). Each item has a minimum score of 1 and a maximum score of 4, and were averaged to create a total score range of 1-4. Higher scores reflect worse outcomes (worse communication). Population: Number analyzed in row differs from overall because this specifically looked at Veteran reports of family communication whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  units on a scale
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 2.42 (0.37) | 2.53 (0.41) | 2.48 (0.39)
Number of Veterans with at least 1 Suicide Attempt [Count of Participants; unit: Participants] — These are the number of Veterans who reported at least one or more behaviors in their lifetime that were coded as "actual suicide attempt" using the C-SSRS criteria. A behavior was considered an "actual suicide attempt" if it was a potentially self-injurious act with any intent to die associated with it. The baseline C-SSRS measured instances of suicidal behavior in the past year, as well as during the participant's lifetime. Population: Number analyzed in row differs from overall because this specifically looked at Veteran suicide attempts whereas overall number includes both Veteran and their dyad partner. Therefore the number analyzed is half the total of each condition.
  Participants
    number analyzed (Participants) | 19 | 20 | 39
    (all) | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Veteran Suicidal Ideation
Description: Suicidality will be measured using the Columbia Suicide Severity Rating Scale. The C-SSRS was used across time points to record level of ideation, lifetime suicide attempts, and recent suicide attempts. The follow-up version of C-SSRS measured suicidal ideation and behavior that had occurred since the last assessment. The scale has inter-rater reliability of .97 and has been used extensively in prospective suicide studies. The scale has a minimum value of 0 and a maximum value of 5. Higher scores mean a worse outcome (more severe ideation).
Time Frame: POST TREATMENT ASSESSMENT- After completing intervention (Range 0.30-7.47 months; Mean=2.84 months from baseline); EXTENDED FOLLOWUP- 3-months after providing follow-up up to 1 year from enrollment (Range 3.10-11.43 months; Mean=6.32 months from baseline)
Population: Some participants lost between baseline and post-treatment follow-up and extended 3 month follow up. These groups specifically refer to Veterans (does not include supporting partners) and therefore include about half of the total participants in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Veterans in SAFER: Veteran participants in the SAFER (intervention) condition
- Veterans in I-SPI: Veterans in the I-SPI (control) condition
Arm/Group | Veterans in SAFER | Veterans in I-SPI
Number analyzed (Participants) | 15 | 15
units on a scale
  Post-Treatment | 1.50 (1.93) | 3.50 (1.43)
  Extended Follow-Up: number analyzed (Participants) | 11 | 14
  Extended Follow-Up | 1.00 (1.31) | 3.38 (2.13)
Statistical Analysis 1: Comparison: Veterans in SAFER vs Veterans in I-SPI; Test type: Superiority; p = .03, Hierarchical Linear Modeling/MLM — All p-values are two-tailed; Hypothesis tested using a dummy code representing group assignment (1=SAFER; 0=I-SPI) in the Level 2 equation for the slope term; Slope = -0.37, Standard Error of Mean 0.17 — Slope represents relative unit change/month between both conditions. Positive slope terms represent relative increases in SAFER compared to I-SPI. Negative slope terms represent relative reductions in SAFER compared to I-SPI

2. Primary Outcome: Supporting Partner Caregiver Burden
Description: Caregiver burden will be evaluated by the Caregiver Burden Inventory (CBI), a 24-item scale assessing caregiver burden in four areas: physical, social, emotional and time dependence burden. Investigators found a large effect size in the pilot multifamily group study on this scale (Cohen's d = 1.03). Items were averaged to create an overall measure of caregiver burden and showed excellent internal consistency in this study (α =.94). CBI scores range from 0 (minimum) to 4 (maximum). Higher scores mean a worse outcome (greater caregiver burden).
Time Frame: as for outcome 1
Population: Some participants lost between baseline and post-treatment follow-up and extended 3-month follow-up. These groups specifically refer to supporting partners (does not include Veterans) and therefore include about half of the total participants in the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Caregivers in SAFER: Caregivers in the SAFER (intervention) condition
- Caregivers in I-SPI: Caregivers in the I-SPI (control) condition
Arm/Group | Caregivers in SAFER | Caregivers in I-SPI
Number analyzed (Participants) | 13 | 13
units on a scale
  Post-Treatment | 1.23 (0.85) | 1.00 (0.86)
  Extended Follow-Up: number analyzed (Participants) | 8 | 13
  Extended Follow-Up | 0.90 (0.59) | 0.72 (0.67)
Statistical Analysis 1: Comparison: Caregivers in SAFER vs Caregivers in I-SPI; Test type: Superiority; p = .69, Hierarchical Linear Modeling/MLM; [statistical method as in outcome 1, analysis 1]; Slope = -0.02, Standard Error of Mean 0.05 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Number of Veterans With at Least 1 Suicide Attempt
Description: These are the number of Veterans who reported at least one or more behaviors coded as "actual suicide attempts" since last visit using the Columbia Suicide Severity Rating Scale (C-SSRS). The follow-up version of C-SSRS measured suicidal ideation and behavior that had occurred since the last assessment. The scale has inter-rater reliability of .97 and has been used extensively in prospective suicide studies. A behavior was considered an "actual suicide attempt" if it was a potentially self-injurious act with any intent to die associated with it.
Time Frame: as for outcome 1
Population: Some participants lost between baseline and post-treatment follow-up and extended 3-month follow-up. These groups specifically refer to Veterans (does not include supporting partners) and therefore include about half of the total participants in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Veterans in SAFER | Veterans in I-SPI
Number analyzed (Participants) | 15 | 15
Participants
  Post-Treatment | 0 | 2
  Extended Follow-Up: number analyzed (Participants) | 11 | 14
  Extended Follow-Up | 0 | 1
Statistical Analysis 1: Comparison: Veterans in SAFER vs Veterans in I-SPI; Test type: Superiority; p = .49, Fisher Exact — All p-values are two-tailed; Compares veterans who reported 1+ attempts at any follow-up wave out of total number of veterans in each group (i.e., 0/19 for SAFER; 2/20 for I-SPI)

4. Secondary Outcome: Veteran Suicide Related Coping
Description: Suicide-related coping will be evaluated by the Stanley Suicide-related Coping Scale (SRCS), a 21-item self-report measure developed by Stanley, Green, Holloway, Brenner & Brown to evaluate appraisal of one's ability to cope with suicidal ideation and urges, as well as ability to use the Safety Plan. Examples of items are: "I am at the mercy of my suicidal thoughts", "I have several things I can do to get through a suicidal crisis". Scores were averaged so that higher scores represent greater confidence and breadth of approaches to coping with suicidal thoughts and feelings (better outcome). SRCS scores have a minimum of 0 and a maximum of 4.
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Veterans in SAFER | Veterans in I-SPI
Number analyzed (Participants) | 15 | 15
units on a scale
  Post-Treatment | 3.15 (0.71) | 2.69 (1.02)
  Extended Follow-Up: number analyzed (Participants) | 11 | 14
  Extended Follow-Up | 3.12 (0.59) | 2.70 (0.86)
Statistical Analysis 1: Comparison: Veterans in SAFER vs Veterans in I-SPI; Test type: Superiority; p = .03, Hierarchical Linear Modeling/MLM; [statistical method as in outcome 1, analysis 1]; Slope = 0.08, Standard Error of Mean 0.04 — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Veteran Thwarted Belongingness
Description: Thwarted belongingness will be evaluated by Interpersonal Needs Questionnaire (INQ-15). The INQ is has demonstrated acceptable internal consistency for thwarted belongingness in this sample (TB) (α =.79). Scores on each subscale were averaged so that higher scores represent a greater degree of their respective constructs. Thwarted belongingness scores range from 1 (minimum) to 6 (maximum). Higher scores mean a worse outcome (decreased feelings of belongingness).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Veterans in SAFER: Veteran participants in the SAFER (treatment) condition
Arm/Group | Veterans in SAFER | Veterans in I-SPI
Number analyzed (Participants) | 15 | 15
units on a scale
  Post-Treatment | 2.85 (1.27) | 3.57 (1.22)
  Extended Follow-Up: number analyzed (Participants) | 11 | 14
  Extended Follow-Up | 3.30 (1.46) | 3.45 (0.95)
Statistical Analysis 1: Comparison: Veterans in SAFER vs Veterans in I-SPI; Test type: Superiority; p = .87, Hierarchical Linear Modeling/MLM; [statistical method as in outcome 1, analysis 1]; Slope = 0.01, Standard Error of Mean 0.07 — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Partner Support of Suicide-Related Coping
Description: We have developed a family counterpart to the Stanley Suicide-related Coping Scale for Veterans that taps family members' appraisal of their ability to participate effectively in Veteran safety planning. Items include, "I recognize the triggers and warning signs for suicidal ideation/urges for my Veteran" and "I know the numbers for the mobile crisis team to contact and nearest hospital or urgent care facility to accompany my Veteran to in a crisis." This measure will be validated against the more general Family Empowerment Scale. Items were rated on a 0 (Strongly Disagree) to 4 (Strongly Agree) scale and were averaged with higher scores indicating greater self-efficacy when supporting the Veteran through suicidal crises (better outcome). Partner SRCS scores range from 0 (minimum) to 4 (maximum).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregivers in SAFER | Caregivers in I-SPI
Number analyzed (Participants) | 13 | 13
units on a scale
  Post-Treatment | 3.65 (0.46) | 3.36 (0.71)
  Extended Follow-Up: number analyzed (Participants) | 8 | 13
  Extended Follow-Up | 3.70 (0.57) | 2.89 (1.4)
Statistical Analysis 1: Comparison: Caregivers in SAFER vs Caregivers in I-SPI; Test type: Superiority; p = .03, Hierarchical Linear Modeling/MLM; [statistical method as in outcome 1, analysis 1]; Slope = 0.17, Standard Error of Mean 0.08 — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Veteran Perceived Burdensomeness
Description: Perceived burdensomeness will be evaluated by Interpersonal Needs Questionnaire (INQ-15). The INQ is has demonstrated excellent internal consistency for Perceived Burdensomeness (PB) (α= .95). Scores on each subscale were averaged so that higher scores represent a greater degree of their respective constructs. Perceived burdensomeness scores range from 1 (minimum) to 6 (maximum). Higher scores mean a worse outcome (greater perceived burdensomeness).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Veterans in SAFER | Veterans in I-SPI
Number analyzed (Participants) | 15 | 15
units on a scale
  Post-Treatment | 2.23 (1.39) | 2.60 (1.68)
  Extended Follow-Up: number analyzed (Participants) | 11 | 14
  Extended Follow-Up | 2.10 (1.63) | 2.86 (1.42)
Statistical Analysis 1: Comparison: Veterans in SAFER vs Veterans in I-SPI; Test type: Superiority; p = .16, Hierarchical Linear Modeling/MLM; [statistical method as in outcome 1, analysis 1]; Slope = -0.12, Standard Error of Mean 0.08 — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Veteran Hopelessness
Description: Veteran hopelessness will be evaluated by the Beck Hopelessness Scale (BHS), a 20-item self-report measure with adequate reliability and validity which has been predictive of suicide in psychiatric inpatients. The BHS measures three aspects of hopelessness: feelings about the future, loss of motivation, and expectations. Items are true-false and are summed to get a total BHS score, ranging from 0 to 20. Higher scores reflect a worse outcome (greater hopelessness).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Veterans in SAFER | Veterans in I-SPI
Number analyzed (Participants) | 15 | 15
units on a scale
  Post-Treatment | 7.40 (6.49) | 11.73 (7.06)
  Extended Follow-Up: number analyzed (Participants) | 11 | 14
  Extended Follow-Up | 9.09 (7.84) | 12.61 (6.70)
Statistical Analysis 1: Comparison: Veterans in SAFER vs Veterans in I-SPI; Test type: Superiority; p = .81, Hierarchical Linear Modeling/MLM — All p-values are two-tailed; [statistical method as in outcome 1, analysis 1]; Slope = .09, Standard Error of Mean .35 — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Veteran Depression
Description: Veteran depression will be evaluated by the widely-used Beck Depression Inventory-II (BDI-II) (Cronbach's = .92). The BDI-II contains 21 items assessing depressive symptoms, each with minimum scores of 0 and maximum scores of 3. Item scores were summed, leading to a total score range of 0-63. Higher scores mean a worse outcome (more severe depressive symptoms).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Veterans in SAFER | Veterans in I-SPI
Number analyzed (Participants) | 15 | 15
units on a scale
  Post-Treatment | 21.20 (16.92) | 29.07 (18.67)
  Extended Follow-Up: number analyzed (Participants) | 11 | 14
  Extended Follow-Up | 18.33 (16.20) | 31.08 (17.67)
Statistical Analysis 1: Comparison: Veterans in SAFER vs Veterans in I-SPI; Test type: Superiority; p = .55, Hierarchical Linear Modeling/MLM — All p-values are two-tailed; [statistical method as in outcome 1, analysis 1]; Slope = -.37, Standard Error of Mean .62 — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Caregiver's Empowerment to Help Veteran
Description: Caregiving self-efficacy/empowerment will be evaluated using the 12-item family subscale from the Family Empowerment Scale. This scale assesses the family's knowledge of mental health services and perceived ability to manage crises, and has demonstrated sensitivity to change in family intervention studies. Each item has a minimum score of 1 and a maximum score of 5, and were averaged to create a total score range of 1-5. Higher scores mean a better outcome (greater empowerment).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Caregivers in SAFER | Caregivers in I-SPI
Number analyzed (Participants) | 13 | 13
units on a scale
  Post-Treatment | 3.71 (0.78) | 3.91 (0.94)
  Extended Follow-Up: number analyzed (Participants) | 8 | 13
  Extended Follow-Up | 3.91 (0.67) | 3.87 (0.86)
Statistical Analysis 1: Comparison: Caregivers in SAFER vs Caregivers in I-SPI; Test type: Superiority; p = .64, Hierarchical Linear Modeling/MLM — All p-values are two-tailed; [statistical method as in outcome 1, analysis 1]; Slope = .02, Standard Error of Mean .05 — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Veteran's Report of Family Problem Solving
Description: Veterans' reports of family problem solving will be evaluated by the 5-item Problem Solving subscale of the Family Assessment Device (FAD). Subscales have acceptable internal consistency (α = .72 to .83). Each item has a minimum score of 1 and a maximum score of 4, and were averaged to create a total score range of 1-4. Higher scores reflect worse outcomes (lower problem solving ability).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Veterans in SAFER | Veterans in I-SPI
Number analyzed (Participants) | 15 | 15
units on a scale
  Post-Treatment | 2.33 (0.86) | 2.23 (0.81)
  Extended Follow-Up: number analyzed (Participants) | 11 | 14
  Extended Follow-Up | 2.36 (0.64) | 2.40 (1.01)
Statistical Analysis 1: Comparison: Veterans in SAFER vs Veterans in I-SPI; Test type: Superiority; p = .62, Hierarchical Linear Modeling/MLM — All p-values are two-tailed; [statistical method as in outcome 1, analysis 1]; Slope = -.02, Standard Error of Mean .04 — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Veteran's Report of Family Communication
Description: Veterans' reports of family communication will be evaluated by the 6-item Communication subscale of the Family Assessment Device (FAD). Subscales have acceptable internal consistency (α = .72 to .83). Each item has a minimum score of 1 and a maximum score of 4, and were averaged to create a total score range of 1-4. Higher scores reflect worse outcomes (worse communication).
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Veterans in SAFER | Veterans in I-SPI
Number analyzed (Participants) | 15 | 15
units on a scale
  Post-Treatment | 2.34 (0.39) | 2.33 (0.54)
  Extended Follow-Up: number analyzed (Participants) | 11 | 14
  Extended Follow-Up | 2.33 (0.28) | 2.27 (0.44)
Statistical Analysis 1: Comparison: Veterans in SAFER vs Veterans in I-SPI; Test type: Superiority; p = .16, Hierarchical Linear Modeling/MLM — All p-values are two-tailed; [statistical method as in outcome 1, analysis 1]; Slope = .04, Standard Error of Mean .03 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 1 year, 8 months
Groups:
- SAFER: Veterans: SAFER: A novel, 4-session intervention to enhance currently mandated VA suicide safety planning by involving family members to support its implementation. Incorporation of education about suicide risk factors and teaching communication skills of active listening and making a positive request will supply Veterans and family members with the knowledge and tools needed to 1) identify potential warning signs, and 2) discuss Veteran ideation or family concerns. SAFER aims to increase family support for the Veteran to directly mitigate Veteran loneliness and sense of being a burden to others.
  Safe Actions for Families to Encourage Recovery: A novel, 4-session intervention to enhance VA suicide safety planning by involving family members to support its implementation.
- I-SPI: Veterans; I-SPI: Caregivers: The comparison condition will be an assessment-only enhanced treatment-as-usual (E-TAU), incorporating update and use of the safety plan, which will then be uploaded to CPRS so the Veterans' primary mental health providers can access.
  Treatment-as-Usual: The comparison condition will be an assessment-only enhanced treatment-as-usual (TAU).
- SAFER: Caregivers: SAFER: A novel, 4-session intervention to enhance currently mandated VA suicide safety planning by involving family members to support its implementation. Incorporation of education about suicide risk factors and teaching communication skills of active listening and making a positive request will supply Veterans and family members with the knowledge and tools needed to 1) identify potential warning signs, and 2) discuss Veteran ideation or family concerns. SAFER aims to increase family support for the Veteran to directly mitigate Veteran loneliness and sense of being a burden to others.
Arm/Group | SAFER: Veterans | I-SPI: Veterans | SAFER: Caregivers | I-SPI: Caregivers
All-Cause Mortality (participants affected / at risk) | 0/19 | 1/20 | 0/19 | 1/20
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/20 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 1/19 | 1/20 | 0/19 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAFER: Veterans (N=19) | I-SPI: Veterans (N=20) | SAFER: Caregivers (N=19) | I-SPI: Caregivers (N=20)
Knee Operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychiatric Hospitalization (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAFER: Veterans (N=19) | I-SPI: Veterans (N=20) | SAFER: Caregivers (N=19) | I-SPI: Caregivers (N=20)
ER for Urination Issue (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ER for Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The proposed evaluation of SAFER has limitations. First, our strategy only targeted moderate risk suicidal Veterans. Second, there was a relatively small sample size of 39 suicidal Veterans and 39 supporting partners. Third, conducting the study in a high density, urban setting may result in different findings than if conducted in a rural setting. Fourth, the study arms were not matched for treatment dosage (SAFER: 4 sessions versus I-SPI: single session).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03034863/Prot_SAP_000.pdf